CLINICAL TRIAL: NCT07061860
Title: Comparative Study of Retention of Mandibular Denture Bases Three-dimensional (3D) Printing Technique and Metal-reinforced Acrylic Resin
Brief Title: To Evaluate the Complete Mandibular Dentures Produced Via 3D Printing in Comparison to Those Constructed From Metal-reinforced Acrylic Resin Regarding Their Retention
Acronym: retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Ayman Fathy Farouk El-Awadi, assistant professor in Prosthodontics Department, Oral and Dental Research Institution, National Research Centre, Cairo, Egypt., National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8887082022
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Edentulous Alveolar Ridge
Keywords: digital denture; retention; metal reinforced denture

STUDY DESIGN:
Intervention Model Description: randomozied controlled parallel double blinding study
Who Masked: Investigator, Outcomes Assessor
Masking Description: blinding to patient and operator in intervention from begining
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complete edentulous patient receive 3D printed denture (Experimental): group 1: 10 patients: Complete dentures constructed from poly-methyl methacrylate resin were used to create the mandibular and maxillary 3D-printed dentures
  Interventions: Device: digital complete denture
- complete edentulous patient receive metal reinforced denture (Active Comparator): group 2: 10 patients: complete denture constructed from metal reinforced acrylic denture
  Interventions: Device: metal reinforced complete denture

INTERVENTIONS:
Device: digital complete denture — different method of denture construction
  Arms: complete edentulous patient receive 3D printed denture
Device: metal reinforced complete denture — different method of denture construction
  Arms: complete edentulous patient receive metal reinforced denture

SUMMARY:
in this study we will construct denture for patient by different way and material one of this denture constructed digitally and the other one constructed in conventional way with metal reinforced. then we will measure the retention of the dentures

DETAILED DESCRIPTION:
the complete denture is constructed for completely edentulous patient. the different technique of construction aim to increase retention of denture to prevent dislodgment during mastication

ELIGIBILITY:
Inclusion Criteria:

* Class I maxillary-mandibular relationship
* well-maintained oral mucosa
* normal salivary flow

Exclusion Criteria:

* smokers patient
* patient had any abnormalities in hard or soft tissues
* severe ridge undercut
* patient received radiation therapy to the head and neck region

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
retention measurement | immediatlly after denture construction
  To assess retention, a digital force gauge (Digital Force Gauge EXTECH 475044) was employed. All of the mandibular dentures were modified to receive a custom-made metal framework consisting of three tubes connected by a hook at the determining geometric center of the denture, two tubes extend 2 cm above the occlusal plane from the retromolar pad region, and one was made at the midline region lingual and below the central incisors. The mandibular denture's polished surface was then joined to the specially constructed custom-made metal framework using self-curing acrylic resin

CONTACTS AND LOCATIONS:
Overall Officials: Ayman F Elawady, Ass prof, Principal Investigator — National research center, cairo, Egypt
Locations (1):
- National Resaerch Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to share

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT07061860/Prot_SAP_000.pdf